CLINICAL TRIAL: NCT02235441
Title: Effects of Chemoradiation and Surgery on Cardiopulmonary Fitness and Tumor Neoplastic Phenotype in Gastrointestinal Malignancies: A Pilot Study
Brief Title: Effects of Chemoradiation and Surgery on Cardiopulmonary Fitness and Tumor Neoplastic Phenotype in Gastrointestinal Malignancies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00055718
Record Dates: First submitted 2014-08-29; First posted 2014-09-10 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pathologically Proven Gastrointestinal Malignancy; Plan of Care Must Include Chemoradiation
Keywords: Gastrointestinal malignancy; Cardiopulmonary fitness; Chemoradiation therapy
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiopulmonary Fitness (Experimental): All eligible subjects will participate in treadmill exercise to measure cardiopulmonary fitness during chemoradiation therapy.
  Interventions: Other: Cardiopulmonary Exercise Test (CPET)

INTERVENTIONS:
Other: Cardiopulmonary Exercise Test (CPET) — All subjects will undergo a maximal cardiopulmonary exercise test and resting metabolic rate study. Prior to the exercise treadmill test, each subject will have a resting ECG and blood pressure to determine whether there are any abnormalities that would contraindicate exercise testing.This exercise test involves exercising on a treadmill to maximal exertion, during which the subject's breathing and oxygen consumption are measured. The subject will wear nose clips to prevent exhaling air through their nose and a mouth piece that will allow all exhaled air to be analyzed through the metabolic cart. The subject's electrocardiogram (ECG), blood pressure, and perceived exertion are monitored throughout the test by trained personnel.
  Other Names: Treadmill exercise

SUMMARY:
There is growing evidence of the integral role of exercise following cancer treatment. Randomized trials show that exercise improves post treatment symptoms and quality of life in breast and prostate cancer patients.Regular exercise reduces cancer specific and all cause mortality for patients with breast, prostate, brain or colorectal cancer. Nearly a 40-50% relative risk reduction in cancer specific death and 20-50% relative risk reduction in all cause mortality have been reported with exercise. At present it is unknown if preclinical pleiotropic effects on tumors through aerobic exercise are clinically relevant. Before launching into further studies of exercise training on changes in tumor hypoxia and response to CRT in rectal cancer patients, it is first important to understand: 1. Whether measures of exercise exposure (i.e., exercise capacity and self-reported exercise behavior) are associated with markers of tumor hypoxia at diagnosis (prior to initiation of CRT) and 2. Whether changes in measures of exercise exposure over the course of CRT are related to changes in tumor hypoxia and response to CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastrointestinal malignancy
2. Plan for chemoradiation
3. At least 18 years old
4. Karnofsky performance status of at least 70% at study entry
5. Ability to read and understand English
6. Signed informed consent prior to initiation of study-related procedures
7. All women of childbearing potential must have a negative serum pregnancy test prior to study entry

Exclusion Criteria:

1. Significant cardiac disease (i.e., left ventricular ejection fraction of <50%, unstable angina, placement of cardiac stents and myocardial infarction within previous 6 months)
2. Contraindications to a cardiopulmonary exercise test as recommended by the American Thoracic Society: (a) acute myocardial infarction (3-5 days), (b) unstable angina, (c) uncontrolled arrhythmias causing symptoms or hemodynamic compromise, (d) syncope, (e) acute endocarditis, (f) acute myocarditis or pericarditis, (g) uncontrolled heart failure, (h) acute pulmonary embolus or pulmonary infarction, (i) thrombosis of lower extremities, (j) suspected dissecting aneurysm, (k) uncontrolled asthma, (l) pulmonary edema, (m) room air desaturation at rest ≤85%, (n) respiratory failure, (o) acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise, (p) mental impairment leading to inability to cooperate, and (q) extensive bone metastases
3. KPS<70%
4. Females who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

PRIMARY OUTCOMES:
Feasibility Composite Score | 36 months
  The primary objective is to determine the feasibility of assessing cardiopulmonary fitness pre and post chemoradiation therapy. This feasibility assessment will be reported as a composite of the following variables: (a) the study can accrue 25 patients in no more than 3 years, (b) at least 18 of these 25 patients adhere to the cardiopulmonary testing pre and post CRT; do not drop out early, and do not have an exercise-related adverse event (i.e., cardiac arrhythmias or myocardial infarction), and (c) no more than 1 patient has an exercise-related adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke Health
Locations (1):
- Joan Cahill, Durham, North Carolina, United States